CLINICAL TRIAL: NCT04432753
Title: Effect of Incidental Findings Information on Lung Cancer Screening Intent: A Randomized Controlled Trial
Brief Title: Effect of Incidental Findings Information on Lung Cancer Screening Intent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: UNC Cecil G. Sheps Center for Health Services Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 19-2709
Record Dates: First submitted 2020-05-28; First posted 2020-06-16 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Neoplasm of Lung; Decision Support Techniques; Mass Screening
Keywords: Incidental Findings
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid with incidental findings information (Experimental): Participants in this arm will view a video decision aid that include information on incidental findings in lung cancer screening.
  Interventions: Behavioral: Lung Cancer Screening Decision Aid with Incidental Findings Information
- Decision aid without incidental findings information (Active Comparator): Participants in this arm will view a video decision aid that does not include information on incidental findings in lung cancer screening.
  Interventions: Behavioral: Lung Cancer Screening Decision Aid without Incidental Findings Information

INTERVENTIONS:
Behavioral: Lung Cancer Screening Decision Aid with Incidental Findings Information — The intervention consists of a previously tested and developed brief lung cancer screening video decision aid with the addition of information on incidental findings for lung cancer screening.
  Arms: Decision aid with incidental findings information
Behavioral: Lung Cancer Screening Decision Aid without Incidental Findings Information — The intervention consists of a previously tested and developed brief lung cancer screening video decision aid that does not include information on incidental findings.
  Arms: Decision aid without incidental findings information

SUMMARY:
This online randomized controlled trial seeks to determine if inclusion of incidental findings information in a lung cancer screening decision aid affects screening intent among screening-eligible individuals. Participants will view either a decision aid with incidental findings information or without and indicate their intent to pursue lung cancer screening.

Hypothesis: Inclusion of incidental findings in a decision aid will decrease intent to screen among participants.

ELIGIBILITY:
Inclusion Criteria:

* 55-80 year old male or female
* Current or former smoker who quit within the last 15 years
* At least 30 pack years of smoking

Exclusion Criteria:

* N/A

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-08-22 (Actual); Study Completion 2020-08-22 (Actual)

PRIMARY OUTCOMES:
Percentage of individuals who plan to pursue lung cancer screening | Day 1
  This will be assessed by a survey item where participants indicate their response to a statement of whether they plan to pursue lung cancer screening, with answer choices being strongly agree, agree, disagree and strongly disagree. Comparison between the intervention and control groups will be made.

SECONDARY OUTCOMES:
Mean score on scale of lung cancer screening knowledge | Day 1
  Lung cancer screening knowledge tested by 6 multiple choice questions on facts of the benefit and harms of screening. The questions will be answered before and after participants watch a lung cancer screening decision aid. Scores will be determined by the number of correct answers for questions.
Mean rating of benefit and harms of screening | Day 1
  Participants will rate (Likert 1-5 scale with 1 being less important and 5 being more important) 6 lung cancer screening benefits and harms on importance to them.
Percentage of Time Lung Cancer Screening Benefit and Harms are ranked first and last | Day 1
  Participants will rank six lung cancer screening benefits and harms.
Mean ranking of benefit and harms of screening | Day 1
  Participants will rank six lung cancer screening benefits and harms.
Percentage of time each lung cancer screening harm is ranked highest of the five potential harms | Day 1
  Participants will rank six lung cancer screening benefits and harms.
Mean ranking of incidental findings attribute | Day 1
  Participants will rank six lung cancer screening benefits and harms, including one on incidental findings. Comparison of mean ranking will be made between the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Clark, MD, Principal Investigator — University of North Carolina, Chapel Hill; Daniel Jonas, MD, MPH, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Clark SD, Reuland DS, Brenner AT, Jonas DE. Effect of Incidental Findings Information on Lung Cancer Screening Intent: a Randomized Controlled Trial. J Gen Intern Med. 2022 Nov;37(14):3676-3683. doi: 10.1007/s11606-022-07409-4. Epub 2022 Feb 2. PMID 35113322